CLINICAL TRIAL: NCT05782114
Title: Efficacy Of Extracorporeal Shockwave Therapy On Ultrasonographic Changes, Pain, Function And Grip Strength In De Quervain Tenosynovitis
Brief Title: Efficacy of Extracorporeal Shockwave Therapy on Ultrasonographic Changes in de Quervain Tenosynovitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Gomaa Mahmoud Ali, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004162
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: De Quervain Disease
Keywords: Extracorporeal Shockwave therapy :ESWT; Ultrasonography US; HandGrip Strenght; De Quervain Tenosynovitis
MeSH Terms: conditions — De Quervain Disease | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Extracorporeal Shockwave therapy &Traditional physical therapy program
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental Group A (Experimental): Extracorporeal Shockwave therapy (four sessions one session per week)
  +Traditional physical therapy program (Instruction to wear Thumb Spica splint, Ultrasound therapy, stretching exercise & strengthening exercise) (two sessions per week for 4 weeks).
  Interventions: Other: Extracorporeal Shockwave therapy; Other: Traditional physical therapy program
- The control Group B (Active Comparator): Traditional physical therapy program (Instruction to wear Thumb Spica splint, Ultrasound therapy, stretching exercise & strengthening exercise) (two sessions per week for 4 weeks).
  Interventions: Other: Traditional physical therapy program

INTERVENTIONS:
Other: Extracorporeal Shockwave therapy — The shockwave will be applied for the experimental group (Group A). The patients will be positioned on a chair, and the hand with the disorder will be placed on a surface with the radio ulnar joint will be in mid position and the thumb will be directed up. will be 1000 impulses with 2 bar pressure at a frequency of 15 Hz on the radial head and focused on the tissue surrounding the maximal pain point.
  Arms: The experimental Group A
Other: Traditional physical therapy program — 1. Instruction to wear Thumb Spica splint:
     The Thumb Spica splint will be used for 4 weeks for both groups of patients.
  2. Ultrasound Therapy:
     Therapeutic Ultrasound parameters will be mode: continuous, duration: 5 minutes, intensity: 1.2watt/cm2 and frequency: 1MHZ.
  3. Stretching exercise:
  1. Self-stretch of the thenar eminence: 2. Opposition stretches: 3. Wrist stretch:
  4) Strengthening exercise:
  1. Resisted exercise for thumb extension:
  2. Resisted exercise for thumb abduction:
  3. Resisted exercise for thumb opposition:
  4. Wrist radial deviation strengthening:
  5. Grip strengthening:
  6. Finger spring:

SUMMARY:
The current study will be conducted to explore the efficacy of ESWT on ultrasonographic changes, pain intensity level, upper limb function and hand grip strength in patients with de Quervain tenosynovitis.

DETAILED DESCRIPTION:
De Quervain tenosynovitis (DQT) is a painful condition involving the tendons of the abductor pollicis longus (APL) and extensor pollicis brevis (EPB). The pathogenesis is generally defined as a stenosing condition of the first dorsal compartment of the wrist, characterized by thickening of the extensor retinaculum of APL and EPB, which can cause tendon gliding difficulties and impingement between the tendons and their fibrous sheaths.

The prevalence rate of DQT in the general population is 0.5% for males and 1.3% for females, with peak prevalence at the age of 40-60 years. Female prevalence is 6 to 10 times higher than that in men. De Quervain tenosynovitis is a repetitive strain injury consider postures where the thumb is held in abduction and extension to be predisposing factors. De Quervain tenosynovitis incidence increased by virtue of modern life conditions such as excessive computer use and increased use of cellular phones.

However, little research has been carried out to determine the therapeutic effects of ESWT in DQT, and up till now, there is a gap in literature that explore ESWT efficacy on ultrasonographic changes of DQT. So This current study will be conducted to explore the efficacy of ESWT on ultrasonographic changes, pain intensity level, upper limb function and hand grip strength in patients with de Quervain tenosynovitis.

Sixty patients from both genders will be involved in this study and will be randomly subdivided into two equal groups in number. First Group (A) (Experimental Group) will receive radial Extracorporeal Shockwave therapy plus Traditional physical therapy program and the second Group (B) (Control Group): This group will receive Traditional physical therapy program.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years
2. Both genders (males and females).
3. Normal BMI ranges between 18.5:24.9 kg/m2.
4. Patients will be referred from an orthopedist with diagnosis of DQT.
5. Chronic pain more than 2 months.
6. No history of undergoing physiotherapy modalities or corticosterone injection therapies for any reasons during the past month.
7. De Quervain tenosynovitis patients will be diagnosed based on the standard criteria, including pain and tenderness in the lateral wrist and a positive result for the Finkelstein test.

Exclusion Criteria:

1. History of undergoing physiotherapy modalities or corticosterone injection therapies for any reason during the past month.
2. Subjects with other neurological disorders rheumatologic diseases causing wrist pain.
3. Pregnancy.
4. History of fracture or surgery on the hand.
5. Severe trauma, and coagulation disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic Changes: Thickness in tendons: | Up to Four weeks
  Ultrasonography which is a valid and reliable measure to evaluate tendon structural changes including:
  1. Tendon thickness APL & EPB tendons in mm.
  2. Thickness of hypoechoic area in mm.
Ultrasonographic Changes: Color Doppler activity | Up to Four weeks
  Ultrasonography

SECONDARY OUTCOMES:
Pain intensity level assessment : | Up to Four weeks
  VAS will be used by the patient to mark his/her level of pain on visual analogue scale.
Assessment of upper limb function: | Up to Four weeks
  by Q-DASH (The Arabic Quick-DASH questionnaire) is an 11-item self-report questionnaire extracted from the full-length version of the DASH concerning the patient's health status.
Handgrip Strength assessment: | Up to Four weeks
  Baseline hydraulic hand dynamometer Hand grip strength as a measure of functional performance will be measured using the Baseline hydraulic hand dynamometer (Baseline®, Irvington, NY, USA).
Pinch grip Strength assessment: | Up to Four weeks
  The key pinch will be tested with a Baseline hydraulic pinch gauge (Baseline®, Irvington, NY, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma S Amen, Principal Investigator — Profeesor of Basic Science / Faculty of Physical therapy/ Cairo university; Nabil M Ismail, Principal Investigator — Assistant Prof. of Basic Science/ Faculty of Physical therapy/ Cairo university; Doaa A Elimy, Principal Investigator — Lecturer of Basic Science /Faculty of Physical therapy/ Cairo university; Ahmed S Abd El Basset, Principal Investigator — Lecturer of Radiology / Faculty of Medicine/ Beni Suef University
Locations (1):
- Mostafa Gomaa Mahmoud, Cairo, Egypt